CLINICAL TRIAL: NCT02778737
Title: An Innovative Psychosocial Intervention for the Treatment of Chronic Pain Patients and Their Families
Brief Title: Acceptance and Commitment Therapy and Cognitive Behavioral Therapy for Chronic Pain
Acronym: ALGEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cyprus (Other)
Collaborators: University of Crete (Other)
Responsible Party: Principal Investigator, Maria Karekla, Licensed Clinical Psychologist, Assistant Professor, Peer reviewed ACT trainer, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K3_K1_0b
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Pain
Keywords: ACT, CBT, Randomized controlled trial, Chronic Pain
MeSH Terms: conditions — Chronic Pain; Color Vision Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-based intervention (Experimental): The Acceptance and Commitment Therapy + MTAU consists of an unpublished manual developed for the purposes of the project (Karekla et al., 2013). The 8, 90-min weekly group sessions focus in fostering psychological flexibility or the capacity to engage or change behaviors based on what a situation affords and an individual's goals, needs, and desires (Hayes et al., 2004). The ACT protocol involves helping patients to engage in values-based behaviors while remain in contact with pain, especially, when efforts to control or reduce it fail or contribute to suffering.
  Interventions: Behavioral: ACT-based intervention
- CBT-based intervention (Active Comparator): The Cognitive Behavioral group + MTAU consists of an unpublished manual developed by Kalantzi-Azizi & Karademas (2003). It includes 8, 90-min weekly group session and primarily focuses on teaching patients to manage their pain by utilizing various techniques, such as activity pacing, muscle relaxation(i.e., progressive muscle relaxation, diaphragmatic breathing, guided imagery), pain recording, thought challenging, problem solving skills, relapse prevention, etc. The CBT protocol involves helping patients to learn to control their pain and to modify dysfunctional thoughts that accompany it.
  Interventions: Behavioral: CBT-based intervention

INTERVENTIONS:
Behavioral: ACT-based intervention — Treatment sessions will be conducted weekly by two co-therapists in groups of approximately 8-10 participants for 1 ½ hours. Although each session has specific objectives, therapists within the time frame, are encouraged to accommodate participants' discussion or other group dynamic issues that may arise.
  Participants will receive their AP-ACT handbook including outlines of each session, activity plan assignments, and a CD with recorded mindfulness exercises.
  Session highlights and AP-ACT activities relevant to each session will be given at each meeting, so that participants will follow along with the treatment protocol. Individuals missing more than two consecutive sessions will be considered as dropouts.
  Arms: ACT-based intervention
Behavioral: CBT-based intervention — Treatment sessions will be conducted weekly by two co-therapists in groups of approximately 8-10 participants for 1 ½ hours. Although each session has specific objectives, therapists within the time frame, are encouraged to accommodate participants' discussion or other group dynamic issues that may arise.
  Participants will receive their AP-CBT handbook including outlines of each session, activity plan assignments, and a CD with recorded relaxation exercises.
  Session highlights and AP-CBT activities relevant to each session will be given at each meeting, so that participants will follow along with the treatment protocol. Individuals missing more than two consecutive sessions will be considered as dropouts.
  Arms: CBT-based intervention

SUMMARY:
Chronic pain is a long-term condition which is related to a number of negative consequences including reduced productivity at work, increased number of sick leave , depression and emotional difficulties among others. Psychological interventions, particular Cognitive Behavioral therapies (CBT) are deemed effective in reducing the negative consequences following a diagnosis of a chronic pain condition. Though research provides substantial evidence for the CBT effectiveness, not all patients manage to reduce pain intensity or improve their physical and psychosocial functioning. Also, CBT appears with only small effect sizes on variables considered to be core domains in chronic pain. Finally, there are criticism targets on the lack of clear mechanisms underlying the process of change in CBT.

New CBT therapeutic approaches, such as Acceptance and Commitment Therapy (ACT) focus on changing individuals' relation with their inner experiences. They utilize mindfulness and acceptance processes, instead of directly changing or controlling the content of internal experiences, as CBT does. ACT has received support for its effectiveness in chronic pain but there are very few clinical randomized trials to compare it with traditional CBT.

The purpose of this study is to determine whether an ACT-based intervention when compared with a CBT-based intervention designed for chronic pain patients is efficacious in reducing pain interference, pain-related disability, and psychological distress. Also this study aims to examine whether any therapeutic effects result due to the effect of acceptance, for those participating in the ACT group or control appraisal, for those participating in the CBT group. Better knowledge of the mechanism of therapeutic change can help us to recognize which patients can be benefit from which approach.

DETAILED DESCRIPTION:
For more than 30 years cognitive behavior therapy has been the mainstream treatment approach for chronic pain patients and research evidence supporting its effectiveness . Review demonstrate that CBT for chronic pain leads in lowered pain, less emotional distress and pain-related disability, reduced medication use and healthcare utilization, and better improvement in physical and psychosocial functioning. Though CBT for chronic pain is effective, recent evidence suggest that not all patients succeed in lowering pain or improving their physical and psychosocial functioning. Also, research shows only small effects on disability and criticisms targets on the lack of clear mechanisms underlying the process of change in CBT. Researchers argue that the problem with CBT effectiveness lies on its methods. CBT attempts to manage various problems that chronic pain patients face utilizing different methods in combination. This expansion of CBT methods has created concerns among researchers and clinicians as it is not clear what works for whom. More comprehensive and integrated theoretical models encompassing various pain coping responses call for new research that can buffer the CBT expansion.

Following the CBT criticisms, new treatment approaches stemming from the third wave of cognitive behavior therapy abandon traditional approaches to directly change or control the content of internal experiences, and give more emphasis on changing individuals' relation with their inner experience. In doing so, they use mindfulness and acceptance approached along with value-committed actions to produce behavioral changes. One of these approaches, known as Acceptance and Commitment Therapy, has extensively researched in the area of chronic pain and recently the division 12 of the APA listed ACT as an empirically treatment with strong research support for general chronic pain conditions. Indeed, ACT has received amounting evidence in chronic pain and research outcomes demonstrate strong effects on physical and psychosocial disability, mood and daily functioning. Though ACT has received support for its effectiveness in chronic pain, there are yet very few clinical randomized trials to compare it with traditional CBT.

The primary aim of the Algea study is to investigate the efficacy of an ACT-based intervention designed for general chronic pain patients and compare it with a CBT intervention. Specific hypotheses include: (1) ACT will demonstrate improvements in pain indices (pain severity and interference), psychological distress, and quality of life when compared with the CBT group; (2) ACT will present with long-term effects (i.e., 6 months) and patients will report better satisfaction with this treatment than the CBT group; and (3) pain acceptance and values-based actions are considered mechanism of change variables that mediate treatment response in ACT, while control appraisal will mediate treatment response in CBT.

Better knowledge of the differences and similarities of the two CBT approaches (i.e., traditional CBT for chronic pain and ACT) in managing chronic pain can help us formulate treatments that can be tailored to patients needs.

ELIGIBILITY:
Inclusion Criteria:

* Presentation of chronic pain episodes
* Significant impact of the chronic pain condition on quality of life
* Having a medical diagnosis of chronic pain
* Stable medical treatment for at least 2 months
* Reading ability sufficient to comprehend self-monitoring forms as well as competence in the Greek language

Exclusion Criteria:

* An active non pharmacologically-controlled psychotic spectrum condition or manic episode, suicidal ideation/ intent or substance use problems within the 6 months prior to recruitment
* Having a severe medical condition in the present (e.g. cancer)
* No significant cognitive impairment, as assessed using the Mini-mental Status Examination (MMSE).
* Age under 18 or above 70 years
* Receiving any other psychological intervention which is based on CBT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity as assessed with the Greek Brief Pain Inventory (G-BPI) | Change from baseline pain intensity through study completion, an average of 1 year
  is an 11-item measure of intensity and interference of pain in 7 life dimensions: work, mood, activity, sleep, relationships, walking and enjoyment, rated on a scale with 0="no pain" and 10="pain as bad as you can imagine". The G-BPI has shown good reliability, Cronbach's alpha=.80 and sufficient validity with constructs considered theoretically related.

SECONDARY OUTCOMES:
Change in the Quality of life as assessed with the Short Form Health Survey (SF-36; Greek version 1.0; Pappa, Kontodimopoulos & Niakas, 2005) | Change in levels of QoL from baseline through study completion, an average of 1 year
  The SF-36 is a 36 items multipurpose measure assessing physical and mental health indexes. It yields a total score indicating a general health index. SF-36 uses a Likert-type scale and higher scores indicate better overall quality of life. The SF-36 is widely used in clinical studies and evidence across studies indicate that it presents with high validity when compared with theoretically related scales. Also across studies SF-36 yields sufficinet chronbach alpha reliability.
Change in insomnia as assessed with the Athens Insomnia Scale (AIS; Soldatos, Digeos, Paparrigopoulos, 2000) | Change in insomnia from baseline through study completion, an average of 1 year
  The AIS is an 8 item scale assessing difficulty with sleep induction, awakenings during the night, early morning awakening, total sleep time, and overall quality of sleep. It uses a Likert-type scale with items ranging from 0= no problem at all to 3= serious problem. AIS has a long and brief version.The long version utilizes the entire eight-item scale (AIS-8) with a total score ranging from 0 (i.e., absence of any sleep-related problem) to 24 (i.e. the most severe degree of insomnia) and assesses a full range of insomnia symptoms reflecting the disorder as it is described in the ICD-10. The brief five-item version (AIS-5) is limited to the first five items, and yields a total score ranged from 0 to 15. AIS-5 evaluates difficulties with sleep quantity and quality. The AIS (both versions) demonstrates good convergent validity when assessed with theoretically related scales and excellent reliability (a=.89 for the AIS-8 and a=.88 for the AIS-5).
Change in the levels of psychological distress as assessed with the Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) | Changes in the levels of psychological distress from baseline through study completion, an average of 1 year
  HADS is a 14 item questionnaire assessing levels of anxiety and depression symptomatology. Each subscale consists of 7 items rated on a 4-point scale (0-3). Higher scores indicate greater psychological distress. The Greek version presents with high internal consistency (Cronbach's alpha=.88) and sufficient validity when compared with scales considered theoretically related (Michopoulos et al., 2008).

OTHER OUTCOMES:
Changes in the levels of pain acceptance as assessed via the Greek Chronic Pain Acceptance Questionnaire (G-CPAQ; Vasiliou, Karekla, Michaelides, & Kasinopoulos, under review) | Changes in pain acceptance from baseline through study completion, an average of 1 year
  The G-CPAQ assesses pain acceptance and consists of 20 items (long version) of which 8-items comprise the short version. It is rated on a 7-point Likert scale (0 = "never true" to 6 = "always true") and yields a total sum with a range from 0-120. Higher scores denote greater pain acceptance. The G-CPAQ presents with sufficient construct validity when assessed with scales considered theoretically related and appears with high reliability (Cronbach's alpha: Total score = .76; AE =.86; PW = .69 for the G-CPAQ-8).
Changes in avoidance of pain levels as assessed via the Greek version of the Psychological Inflexibility in Pain Scale (G-PIPS-II; Vasiliou, Karekla, Michaelides, & Kasinopoulos, in preparation; Wicksell, Lekander, Sorjonen & Olsson, 2010) | Changes in pain avoidance from baseline through study completion, an average of 1 year
  The G-PIPS-II contains 12 items assessing pain-related avoidance. Items are rated on a 7-point Likert-type scale, with 1="never true" and 7="always true". Higher scores indicate higher avoidance of pain. The scale shows good psychometric properties (Wicksell et al. 2010) with high internal consistency (Cronbach's a=.88) and validity with associated constructs in its Greek version. The PIPS-II scale is frequently used a a coping with pain scale assessing pain avoidance.
Changes in experiential avoidance as assessed via the Acceptance and Action Questionnaire- Greek version (AAQ-II; Karekla & Michaelides, under review) | Changes in experiential avoidance from baseline through study completion, an average of 1 year
  The Acceptance and Action Questionnaire- Greek version is a 7-item measure of experiential avoidance or an individual efforts to systematically avoid or control unwanted internal experiences such as thoughts, emotions, bodily sensations etc (Hayes et al, 2004). It uses a Likert-type scale ranging from 1="never true" to 7="always true". Higher scores indicate greater experiential avoidance. The measure demonstrated good psychometric properties (Cronbach's alpha=.83) and a unidimensional factor structure in its original version (Bond et al., 2011). Also, validation of the AAQ-II in the Greek language present with similar with its english counterpart psychometric properties (alpha=.92).
Changes in mindfulness as assessed via the Cognitive Affective Mindfulness Scale-Revised (CAMS-R; Feldman, Hayes, Kumar, Greeson, & Laurenceau, 2007) | Changes in mindfulness levels from baseline through study completion, an average of 1 year
  The CAMS-R is a 12 item questionnaire assessing mindfulness. Items are rated on a 4-point Likert scale from 1="rarely" to 4="almost always". Cronbach's alpha ranges from .74 to .77 (Feldman et al., 2007). CAMS-R presents with high reliability (a = .81) and sufficient construct validity as assessed with theoretically related constructs. A Greek version appears with similar to its English counterpart unitary factor structure, high reliability (a =.88) and sufficient construct validity with other theoretically-related scales.
Changes in goal-directed behaviors as assessed via the Committed Action Questionnaire (CAQ; McCracken et al., 2014) | Changes in goal-directed behaviors from baseline through study completion, an average of 1 year
  CAQ is an 8-item scale assesses goals- directed behaviors (McCracken, 2014). Items are ranged from 0 = never true to 6 = always true, and higher scores denote higher committed actions. CAQ presents with high internal consistency reliability (a = .87) and sufficient validity with other related instruments, including pain acceptance, depression, and functioning (McCracken et al., 2014).
Changes in living composite values as assessed via the Valued Living Questionnaire (VLQ; Wilson, Sandoz, Kitchens, & Roberts, 2010) | Changes in living composite values levels from baseline through study completion, an average of 1 year
  VLQ assesses individuals' values and the degree to which they live consistently with these values in their everyday life. It consists of two factors (i.e. importance and consistency). Respondents are asked to rate 10 areas of life (e.g. family, relationships, work, education etc.) on a scale of 1= the worst level of important/ consistency in each domain and 10= the highest level of importance/ consistency in each domain. The living composite which represents the degree to which a person lives and behaves in accordance to chosen values, is calculated by summing the importance and consistency responses for each item (Wilson, 2008). Preliminary studies demonstrate that the VLQ has adequate reliability a = .74 (Wilson et al., 2010). Reliability of the Greek version of the VLQ is high for both factors (Importance: a = .81; Consistency: a =.87) and the living composite total score (a =.89; Stavrinaki, Siamata, Vasiliou, Karekla & Kasinopoulos, 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Crete, Rethymno, Crete, Greece

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request and after the sponsor's permission.